CLINICAL TRIAL: NCT00252681
Title: Surgery for Necrotizing Enterocolitis in Human Infants: A Randomized Trial
Brief Title: Comparison of Two Surgical Treatments for Necrotizing Enterocolitis in Human Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD038462 (NIH); Gen Clin Res Ctr #M01-RR00125
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-11

CONDITIONS: Necrotizing Enterocolitis
Keywords: randomized; controlled; trial; necrotizing; enterocolitis; premature; infants; laparotomy; peritoneal; drainage
MeSH Terms: conditions — Enterocolitis, Necrotizing; Enterocolitis; Premature Birth | interventions — Laparotomy

INTERVENTIONS:
Procedure: laparotomy
Procedure: primary peritoneal drainage

SUMMARY:
The primary purpose of this study is to compare two surgical treatments for perforated necrotizing enterocolitis in very low birth weight babies.

DETAILED DESCRIPTION:
This is a multi-center randomized clinical trial comparing laparotomy vs peritoneal drainage for perforated Necrotizing Enterocolitis. The current literature does not allow an objective comparison between these two methods. A recent comprehensive meta-analysis of all published and much unpublished data regarding the use of these procedures in the treatment of perforated NEC revealed that the degree of bias in assignment to treatment precluded an adequate determination as to the best treatment. The conclusion that only a randomized clinical trial would answer this question has led to this multi-center effort. The relative infrequency of the disease at any one neonatal center has necessitated enrollment of patients at many centers.

Comparison: Premature neonates weighing less than 1500 grams at birth who develop perforated necrotizing enterocolitis are randomized within two birth weight blocks (<1000 gms and 1000 - 1499 gms) for treatment with either laparotomy or primary peritoneal drainage. Daily postoperative clinical care is kept uniform between the two groups by means of a critical care pathway. The primary outcome variable is mortality, i.e. death within 90 days of intervention. The main secondary outcome is short bowel syndrome - defined as the need for chronic parenteral nutrition greater than 3 months following operation.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight less than 1500 grams
* Gestational age 24 -33 weeks
* Diagnosed with necrotizing enterocolitis based on Bell stage II or greater
* Bowel perforation as evidenced by free intraperitoneal air seen on abdominal radiograph, stool, bile, or pus found at paracentesis or clinical evidence of perforation in the joint opinion of the attending surgeon and neonatologist.

Exclusion Criteria:

* Bilateral Grade IV intraventricular hemorrhage
* Previous abdominal surgery
* Evidence of gastrointestinal anomaly (i.e. atresia, malrotation etc.)

Ages: 0 Years to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130
Dates: Start 1999-07; Study Completion 2005-06

PRIMARY OUTCOMES:
The primary outcome variable is operative mortality, i.e. death within 90 days of intervention.

SECONDARY OUTCOMES:
The secondary outcome is short bowel syndrome - defined as the need for chronic parenteral nutrition greater than 3 months following operation.

CONTACTS AND LOCATIONS:
Overall Officials: R. Lawrence Moss, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine Section of Pediatric Surgery, New Haven, Connecticut, United States

REFERENCES:
- [Result] Moss RL, Dimmitt RA, Barnhart DC, Sylvester KG, Brown RL, Powell DM, Islam S, Langer JC, Sato TT, Brandt ML, Lee H, Blakely ML, Lazar EL, Hirschl RB, Kenney BD, Hackam DJ, Zelterman D, Silverman BL. Laparotomy versus peritoneal drainage for necrotizing enterocolitis and perforation. N Engl J Med. 2006 May 25;354(21):2225-34. doi: 10.1056/NEJMoa054605. PMID 16723614